CLINICAL TRIAL: NCT07184151
Title: Evaluation of Guided Endodontic Microsurgery and Two Different Retrograde Filling Materials:A Randomized Clinical Trial
Brief Title: Evaluation of Guided Endodontic Microsurgery and Two Different Retrograde Filling Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mohamed fouad el marakby, PHD Candidate at the Faculty of Dentistry, Suez Canal University, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (REC) (379/ 2021)
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Endodontic Re-treatment Failure
Keywords: MTA; Well root putty; guided endodontic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- microsurgical apicoectomy without guide+MTA (Active Comparator)
  Interventions: Drug: MTA retrograde filling
- microsurgical apicoectomy without guide+well root putty ( premixed bioceramic putty) retrograde fil (Experimental)
  Interventions: Drug: well root putty ( premixed bioceramic putty) retrograde filling
- microsurgical apicoectomy with guide+MTA (Experimental)
  Interventions: Drug: MTA retrograde filling
- microsurgical apicoectomy with guide+well root putty ( premixed bioceramic putty) retrograde fil (Experimental)
  Interventions: Drug: well root putty ( premixed bioceramic putty) retrograde filling

INTERVENTIONS:
Drug: well root putty ( premixed bioceramic putty) retrograde filling — well root putty ( premixed bioceramic putty) retrograde filling
  Arms: microsurgical apicoectomy with guide+well root putty ( premixed bioceramic putty) retrograde fil; microsurgical apicoectomy without guide+well root putty ( premixed bioceramic putty) retrograde fil
Drug: MTA retrograde filling — MTA retrograde filling
  Arms: microsurgical apicoectomy with guide+MTA; microsurgical apicoectomy without guide+MTA

SUMMARY:
The aim of this study was to evaluate the effect of guided endodontic microsurgical root end resection on bone healing compared to nonguided microsurgery using two different retrograde filling material (Well root putty, MTA) by cone-beam computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Tooth is restorable pocket depth is less than 4mm and mobility in its normal limit ( less than 1mm)
* Persisting or emerging disease following root-canal treatment when root canal re-treatment is inappropriate.
* Tooth with acceptable endodontic treatment and have a new post and crown restoration, but have a persistent or enlarging periapical lesion ( size less than 10 mm)
* Obstructed canal (the obstruction proved not to be removable, by passed and the risk of damage was too great).
* Extruded material or instrument with clinical or radiological findings of apical periodontitis and/or symptoms are present.

Exclusion Criteria:

* Non restorable tooth
* Contraindicating medical condition ( severe systemic condition and psychological condition)
* Anatomical contra indication
* Poor general oral status and supporting periodontal tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Operating time | perioperative
  The operating time was measured from the beginning of osteotomy to the end of retrograde filling procedure

SECONDARY OUTCOMES:
Change in bone density measurement over time | 1 week, 6 months
Pain "Numerical Rating Scale (NRS)" | first day , 1 week
  Pain was categorized into four categorical scores: (1) none [score 0], (2) mild [score from 1-3], (3) moderate [score from 4-6], (4) severe [score from 7-10
Change in Linear measurements over time | baseline and 6 months
  The evaluator located the slice on CBCT that will appear to demonstrate the largest size of the lesion and made a measurement of the lesion at what appeared to be the widest dimension. A second measurement of the widest dimension will be then made at 90 degrees to this initial measurement. These measurements will be made from a bone landmark to another bone landmark. These measurements will be performed in two planes for each lesion.
Bone healing assessment | baseline and at 6 months
  For analysis of periapical radiographic healing, CBCT scans were oriented in the buccolingual plane along the longitudinal axis of the treated roots. The observers rated the radiographic healing based on the parameters described recently by von Arx et al. (2016) in. Healing was categorized and scored as follows: 1. Fully healed (score 2) , Partially healed (score 1) and Not healed (score 0)
Change in volumetric measurement over time | 1 week, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided